CLINICAL TRIAL: NCT03692637
Title: Clinical Study on the Safety and Efficacy of Anti-Mesothelin Car NK Cells With Epithelial Ovarian Cancer
Brief Title: Study of Anti-Mesothelin Car NK Cells in Epithelial Ovarian Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Allife Medical Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mesothelin Car NK-HNRM-01
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-09

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-Mesothelin Car NK Cells (Experimental): Total dose of 0.5-3 million /kg cells will be administered at day0
  Interventions: Biological: anti-Mesothelin Car NK Cells

INTERVENTIONS:
Biological: anti-Mesothelin Car NK Cells — anti-Mesothelin Car NK Cells injection

SUMMARY:
This is a single centre、single arm、open-label，to investigate the safety and efficacy of anti-Mesothelin Car NK Cells With Epithelial ovarian cancer

DETAILED DESCRIPTION:
Ovarian cancer ranks second in gynecologic malignancies, but mortality ranks first. It is one of the most serious malignant tumors that threaten women's lives. It is urgent to explore new treatment methods, such as introduction. Tumor immunotherapy strategies to improve treatment outcomes and patient quality of life. Car is a group of fusion proteins composed of multiple parts, including antigen recognition region, transmembrane region, and NK cell stimulation region. NK cells are naive immune cells that are not restricted by MHI and can be activated without additional co-stimulatory regions. After activation, granulin-B and γ-interferon are released, thereby inducing apoptosis of tumor cells and lysis of tumor cells. The study will follow a 3 + 3 design of dose- escalating cohorts. After a patient enrolls, leukapheresis will be performed to obtain peripheral blood mononuclearcells which will be sent to a manufacturing site to produce anti-Mesothelin Car NK cells. The cells will then be returned to the investigational site and, after a standard chemotherapy based conditioning regimen, will be administered to the patient. Treated patients will undergo serial measurements of safety, tolerability and response.

ELIGIBILITY:
Inclusion Criteria:

1. Mesothelin-positive patients with stage II-IV epithelial ovarian cancer.（Mesothelin expression ≥50% of tumor cells）（Patients with recurrence are not excluded）
2. Male or female, 18 to 70 years old (including 18 and 70 years old)
3. The excepted survival ≥ 6 months,Karnofsky activity function status score ≥ 60 points
4. there are measurable lesions according to the RECIST 1.1 standard.
5. Bone marrow function (blood routine) satisfies: the number of neutrophils > 1×109/L platelet > 7.5×109/L; hemoglobin > 90 g/L; total bilirubin < 2.0 mg/dL; creatinine < 1.5 times the upper limit; albumin < 2 g/L; ALT or AST < 5 times the upper limit; creatinine clearance rateby Cockcroft-Gault formula< 40 mL/min
6. Coagulation parameters: INR ≤ 1.5, PTT < 1.2 times the upper limt
7. Patients did not receive any chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs PD-1, PDL-1) or other anticancer treatment 2-4 weeks before admission, and the treatment-related toxicity reaction ≤1 level prior to enrollment（except low toxicity lose hair for example）
8. Venous channel is unobstructed, which can meet the needs of intravenous drip
9. HIV test was negative; HBV and HCV were negative
10. Voluntary informed consent is given, agree to follow the trial treatment and visit plan

Exclusion Criteria:

1. Patients with hypertension (> 160/95 mmHg) are uncontrollable; coronary heart disease and angina pectoris are unstable (Canadian Cardiovascular Association Level II and above), or recurrent within 6 months
2. Patients suffer from concurrent or central nervous system diseases
3. Patients with severe autoimmune diseases or immunodeficiency diseases
4. Patient's lung function has the following abnormalities: FEV (forced expiratory volume), < 30%; DLCO (diffusing capacity of lung for carbon monoxide) < 30%; oxygen saturation < 90%
5. Patients treated with other immune cellular products (DC, CIK, T, NK, and Car T products with CD19 or other targets)
6. Patients with Severe liver and kidney dysfunction
7. Patients with Severe bacterial and viral infections
8. Patients are pregnant or nursing
9. Patients used corticosteroids within 4 weeks prior to enrollment(except patients with inhaled hormone)
10. Patients participated in other clinical trials within 30 days.
11. Patients had other conditions that were not appropriate for the group determined by the researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v4.0 | Day 3-Year 2 after injection
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events that are possibly, likely, or definitely related to study treatment